CLINICAL TRIAL: NCT03726424
Title: The Clinical Outcome and Prognosis of Patients With Different Pathogenic Mutations of Hypertrophic Cardiomyopathy
Brief Title: Outcome of Different Pathogenic Mutations in Hypertrophic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof., Tongji Hospital
Other Study IDs: PPOHPM
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: pathogenic mutations; clinical phenotype; prognosis
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mutation: patients carrying one or more specific pathogenic mutations
- control: patients not carrying the pathogenic mutation(s)

SUMMARY:
This is a prospective, single-center study to assess clinical phenotype and prognosis of different pathogenic mutations in Chinese patients with hypertrophic cardiomyopathy. Patients with hypertrophic cardiomyopathy were consecutively recruited, and then DNA samples were extracted from peripheral blood. Targeted sequencing of 142 genes was performed to obtain variants associated with hypertrophic cardiomyopathy. Patients will undergo face-to-face interviews, phone calls, or/and chart reviews at 6 months, 12 months, 24 months, 36 months, 48 months and 60 months for data collection of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults: a wall thickness ≥15 mm in one or more LV myocardial segments-as measured by any imaging technique (echocardiography, cardiac magnetic resonance imaging (CMR) or computed tomography (CT))-that is not explained solely by loading conditions;
* 2. Children: an LV wall thickness more than two standard deviations greater than the predicted mean (z-scored>2, where a z-score is defined as the number of standard deviations from the population mean);
* 3. Relatives: the first-degree relatives of patients with unequivocal disease (LVH ≥15 mm) is based on the presence of otherwise unexplained increased LV wall thickness ≥13 mm in one or more LV myocardial segments, as measured using any cardiac imaging technique [echocardiography, cardiac magnetic resonance (CMR) or CT].

Exclusion Criteria:

* 1. Patients with severe valvular disease, aortic stenosis, congenital heart disease, hypertensive heart disease, diabetic cardiomyopathy, or other cardiovascular or systemic diseases that may cause ventricular hypertrophy;
* 2. Patients who had participated in any clinical trial during the first 3 months;
* 3. Previous history of cancer or tumor, or pathological examination confirmed precancerous lesions (such as breast ductal carcinoma in situ, or atypical hyperplasia of the cervix);
* 4. Patients refused to comply with the requirements of this study to complete the research work.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hypertrophic cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-02-25 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality | up to 60 months
  Death from cardiovascular disease which includes coronary artery diseases, stroke, heart failure, hypertensive heart disease, rheumatic heart disease, cardiomyopathy, heart arrhythmia, congenital heart disease, valvular heart disease, carditis, aortic aneurysms, peripheral artery disease, thromboembolic disease, and venous thrombosis
Rate of heart transplantation | up to 60 months
  Heart transplantation is a surgical transplant procedure performed on patients with end-stage heart failure or severe coronary artery disease when other medical or surgical treatments have failed
Rate of nonfatal stroke | up to 60 months
Rate of nonfatal myocardial infarction | up to 60 months

SECONDARY OUTCOMES:
All-cause mortality | up to 60 months
Readmission rate for cardiovascular diseases | up to 60 months
Recurrence rate of heart failure | up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Dao Wen Wang, Doctor, Study Chair — Tongji Hospital,Wuhan, Hubei, China, 430030
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China